CLINICAL TRIAL: NCT03678272
Title: Comparative Study of Inguinodynia After Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Dr. Antonio Arroyo, Head of General surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HGUE-UP-13-01
Record Dates: First submitted 2017-01-30; First posted 2018-09-19 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Inguinal Hernia; Inguinal Hernia Repair; Open Inguinal Hernia
Keywords: Inguinal hernia; Chronic postoperative inguinal pain; Glue mesh; Suture mesh
MeSH Terms: conditions — Hernia, Inguinal | interventions — Herniorrhaphy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HERNIOPLASTY WITH PANAVALE MESH (Active Comparator): Preformed polypropylene mesh.
  Interventions: Procedure: HERNIOPLASTY WITH PANAVALE MESH
- HERNIOPLASTY WITH PARIETEX PROGRIP MESH (Active Comparator): Mesh consisting of mono lament polyester with a resorbable polylactic acid (PLA) microgrip technology.
  Interventions: Procedure: HERNIOPLASTY WITH PARIETEX PROGRIP MESH
- HERNIOPLASTY WITH ADHESIX MESH (Active Comparator): Self-adhesive mesh.
  Interventions: Procedure: HERNIOPLASTY WITH ADHESIX MESH
- HERNIOPLASTY WITH TIMESH MESH (Active Comparator): Titaniumized polypropylene mesh.
  Interventions: Procedure: HERNIOPLASTY WITH TIMESH MESH

INTERVENTIONS:
Procedure: HERNIOPLASTY WITH PANAVALE MESH — Polypropylene mesh fixed with 3 points. Preformed polypropylene mesh will be used by fixing it with one point to the pubis, another to the inguinal ligament and another to the joint tendon.
  Other Names: Coated Vicryl (poliglactin 910) Suture 2-0 ( Ethicon)
  Arms: HERNIOPLASTY WITH PANAVALE MESH
Procedure: HERNIOPLASTY WITH PARIETEX PROGRIP MESH — Preformed polypropylene mesh will be used which presents a self adhesive system not based on glue, but on the arrangement of the fibers of the mesh as "hooks", and to which we will give a single point to the pubis.
  Other Names: Coated Vicryl (poliglactin 910) Suture 2-0 ( Ethicon)
  Arms: HERNIOPLASTY WITH PARIETEX PROGRIP MESH
Procedure: HERNIOPLASTY WITH ADHESIX MESH — It will use a self-adhesive mesh without giving points to fix this one, since it is a mesh that integrates the glue.
  Arms: HERNIOPLASTY WITH ADHESIX MESH
Procedure: HERNIOPLASTY WITH TIMESH MESH — Titaniumized polypropylene mesh will be used without fixing points, since liquid cyanoacrylate (Ifabond) will be used to fix it.
  Other Names: Ifabond Synthetic Surgical Adhesive 1,5 ml (Péters Surgical)
  Arms: HERNIOPLASTY WITH TIMESH MESH

SUMMARY:
To evaluate the postoperative pain and the relapse after the repair of the inguinal hernia by Lichtenstein technique with four different mesh types with different types of fixation in patients undergoing major ambulatory surgery.

DETAILED DESCRIPTION:
Since the widespread use of meshes in the repair of inguinal hernia, recurrence rates have acceptable values, so, today, the focus is on trying to decrease chronic pain after hernioplasty. Chronic postoperative inguinal pain (CPIP) is an important clinical problem, which can significantly influence the quality of life of the patient. Different studies have published CPIP rates from 9.7% to 51.6%.

The reasons for CPIP are unclear; Lesion and entrapment of the nerves, the type of mesh used, and the fixation material of this has been related to the causes of inguinodynia.

CPIP can be divided into neuropathic pain and non-neuropathic pain. According to the International Association for the Study of Pain (IASP), neuropathic pain is caused by the primary lesion or nerve dysfunction, causing burn-like pain that radiates through the area innervated by the injured nerve, intensifying the nerve with light touch. The causes of this type of pain are the entrapment of the nerve by the mesh or sutures or by the formation of neuromas associated with the partial or complete transection of the nerve. The nerves that run through the inguinal region and are therefore susceptible to injury when the anterior approach is the ilioinguinal nerve, the genitofemoral genital branch, and the iliohypogastric nerve.

Neuropathic pain may occur immediately after surgery, but may also occur months or years after surgery.

Non-neuropathic or nociceptive pain is caused by the activation of mediators of inflammation due to the continuous inflammatory reaction that occurs around the mesh. According to Amid, nociceptive pain is caused by the mechanical pressure of the mesh over adjacent tissue, including the vas deferens and nerves. This type of pain is acute and stabbing and is aggravated by intense exercise.

In conclusion, the use of foreign materials in hernia surgery may induce intense inflammation that can result in chronic pain.

The hypothesis of our work is that: "The use of glue-attached meshes (self-adhesive) compared to those fixed with suture present lower rates of post-hernioplasty pain".

ELIGIBILITY:
Inclusion Criteria:

* Age: over 18 years
* Patients undergoing INGUINAL HERNIA surgery on a scheduled basis in surgery without hospitalization.
* Sign informed consent.
* ASA I-II.
* Inguinal hernia.
* Unilateral or bilateral hernia.
* Lichtenstein hernia repair technique

Exclusion Criteria:

* Patients with ASA III-IV.
* Psychiatric disorders.
* Pregnant or breastfeeding.
* Non-acceptance of informed consent.
* No acceptance or inability to follow a follow-up protocol.
* Any hernia repair technique other than Lichtenstein.
* Recurrent inguinal hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2013-04; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pain to the month. | One month.
  Pain measured by visual analog scale. The pain will be measured one month after surgery.
Pain to the sixth month | Six months.
  Pain measured by visual analog scale. The pain will be measured after the sixth month of surgery.
Pain a year | One year.
  Pain measured by visual analog scale. Pain will be measured after the year of surgery.

SECONDARY OUTCOMES:
Recurrence | One year.
  Recurrence is measured by physical examination by a surgeon outside the study. If there are doubts, it is confirmed or discarded by ultrasound of the operated inguinal region.
Surgical time. | Intraoperative
  Duration of surgery from the incision to the closure of the skin. Time measured in minutes.
Hypoaesthesia to the month. | One month.
  Hypoesthesia is defined as a decrease in sensitivity in the operated area and / or that can extend to the skin of the corresponding scrotum, labia majora and Scarpa triangle. Hypoaesthesia will be measured one month after surgery by physical examination.
Hypoesthesia at the sixth month. | Six months.
  Hypoesthesia is defined as a decrease in sensitivity in the operated area and / or that can extend to the skin of the corresponding scrotum, labia majora and Scarpa triangle. Hypoesthesia will be measured at the sixth month after surgery by physical examination.
Hypoesthesia at one year. | One year.
  Hypoesthesia is defined as a decrease in sensitivity in the operated area and / or that can extend to the skin of the corresponding scrotum, labia majora and Scarpa triangle. Hypoaesthesia will be measured one year after surgery by physical examination.
Post-surgery complication. | One month.
  Postoperative complications are recorded after the first month of surgery. They are local complications such as hematoma, seroma, wound dehiscence, wound infection.